CLINICAL TRIAL: NCT03359798
Title: The Effect of a Counseling Intervention on Post-cesarean Section Narcotic Use: a Randomized Controlled Trial
Brief Title: RCT of Counseling Intervention on Post-op Opiate Use
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in practice patterns
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Julian N Robinson, Chief of Obstetrics, Associate Professor of Obstetrics and Gynecology, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017P000792
Record Dates: First submitted 2017-11-21; First posted 2017-12-02 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Post-operative Pain; Opioid Use; Cesarean Section
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Narcotic counseling script (Experimental): Study participants will be read a script regarding post-cesarean section narcotic use.
  Interventions: Behavioral: Narcotic counseling script
- Post-partum depression counseling script (Sham Comparator): Study participants will be read a script of the same length, and much of the same wording as the experimental script. However, this script's content is focused on post-partum depression.
  Interventions: Behavioral: Post-partum depression counseling script

INTERVENTIONS:
Behavioral: Narcotic counseling script — Script regarding post-cesarean section narcotic use
  Arms: Narcotic counseling script
Behavioral: Post-partum depression counseling script — Study participants will be read a script of the same length, and much of the same wording as the experimental script. However, this script's content is focused on post-partum depression.
  Arms: Post-partum depression counseling script

SUMMARY:
This study is a randomized controlled trial to investigate the effect of a simple counseling intervention on post-operative narcotic requirements, with the hypothesis that women receiving this intervention will use fewer narcotics for pain management following cesarean section.

DETAILED DESCRIPTION:
All women undergoing scheduled cesarean section at Brigham and Women's Hospital who meet eligibility for the study will be approached in the pre-operative area on the Labor and Delivery floor prior to her scheduled cesarean section. For eligible patients interested in participation, consent will be obtained, and the participant will be randomized to receive either an intervention script containing counseling about post-op narcotic use, or the control script containing information regarding post-partum depression. This script will then be read to the participant in the pre-operative area prior to her scheduled cesarean section.

Two types of data will then be collected: inpatient data, and outpatient data. Regarding inpatient data, study investigators will collect information from the electronic medical record about the quantity of narcotics used in the hospital, pain scores while in the hospital, and demographic information. In terms of outpatient data, study investigators will contact participants at 2 weeks and 6 weeks post-partum with questions from the Edinburgh post-partum depression scale score and the WHOQOL-BREF scale score, along with questions regarding their narcotic use at home. Specifically, participants will be asked during the informed consent process whether they agree to 1) receive an email with a brief online survey at 2 weeks post-partum, and 2) receive a follow-up phone call within the week after the email survey was sent if survey responses are not received, 3) receive a second email with a brief online survey at 6 weeks post-partum, 4) receive a follow-up phone call within the week after the second email survey was sent if survey responses are not received. Surveys will be emailed to participants using the Partner's REDCap service that is located behind the Partner's firewall. Investigators will also mine information about each participant's narcotic use from the MassPAT prescription monitoring database.

The endpoint of the study will be enrollment of our desired sample size.

ELIGIBILITY:
Inclusion Criteria:

* Delivery by scheduled cesarean section at Brigham and Women's Hospital

Exclusion Criteria:

* Answer "yes" to the question: "Has any provider talked to you this pregnancy about medications for pain control after your c-section?"
* History of opiate abuse
* Use of chronic opiates, benzodiazepines or gabapentin
* History of chronic pain
* Cesarean hysterectomy
* Vertical skin incision
* Myomectomy at the time of cesarean section
* Non English-speaking
* Patient of the investigator performing the recruitment

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
quantity of narcotics used in-hospital | 4 days

SECONDARY OUTCOMES:
quantity acetaminophen used in-hospital | 4 days
quantity ibuprofen used in-hospital | 4 days
quantity ketorolac used in-hospital | 4 days
pain scale in-hospital | 1 day, 4 days
narcotic prescription filled after discharge | 2 weeks
quantity of narcotics taken after discharge | 2 weeks
Edinburgh post-partum depression score | 2 weeks and 6 weeks

REFERENCES:
- [Derived] Zimpel SA, Torloni MR, Porfirio GJ, Flumignan RL, da Silva EM. Complementary and alternative therapies for post-caesarean pain. Cochrane Database Syst Rev. 2020 Sep 1;9(9):CD011216. doi: 10.1002/14651858.CD011216.pub2. PMID 32871021